CLINICAL TRIAL: NCT06847880
Title: The Potential Effect of the Local Administration of Vitamins C and E on Orthodontic Treatment: a Randomized Clinical Trial
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Ayat M. Hussein, Principal Investigator, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1014425
Record Dates: First submitted 2025-02-01; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Pain Perception; Root Resorption; Rate of Orthodontic Tooth Movement; Biomarkers
Keywords: Orthodontic tooth movement; Root resorption; RANKL; Tooth alignment; Vitamin C; Vitamin E; Pain perception; Osteoprotegerin; RUNX2
MeSH Terms: conditions — Root Resorption | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: This multicenter, prospective, randomized clinical trial follows a parallel-group design (1:1:1) with single blinding. Patients and operators are blinded, but the investigator (A.M.H.) is not. Participants are randomly assigned to one of three groups: (1) Control (saline injection), (2) Vitamin C (ascorbic acid injection), or (3) Vitamin E (alpha-tocopherol injection). Randomization uses a computer-based generator with stratification, and allocation is concealed in sealed containers. Orthodontic tooth movement, root resorption, pain perception, and biomarker levels will be measured at baseline and every four weeks up to 24 weeks. Vitamin injections are administered biweekly for six months (the supposed end date of leveling and alignment stage).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: No additional parties are masked in this clinical trial beyond the participant, care provider, and outcomes assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1: Vitamin C Treatment (Experimental): This arm involves participants receiving Vitamin C to assess its effect on orthodontic tooth movement and crowding relief. The treatment aims to evaluate how Vitamin C influences the rate of tooth movement, as measured by Little's Irregularity Index (LII) over 24 weeks (the supposed end date of leveling and alignment stage).
  Interventions: Drug: 1: Vitamin C Supplementation
- Vitamin E Treatment (Experimental): Participants in this arm will receive Vitamin E to evaluate its effect on orthodontic tooth movement. The aim is to compare the efficacy of Vitamin E to Vitamin C and the saline control in terms of crowding relief and tooth alignment, measured using LII over a 24-week period (the supposed end date of leveling and alignment stage).
  Interventions: Drug: Vitamin E Supplementation
- Arm 3: Saline Control (Placebo Comparator): This arm serves as the control group, where participants receive saline injections. The primary aim is to assess how saline compares with Vitamin C and Vitamin E treatments in terms of the rate of orthodontic tooth movement and crowding relief as measured by LII.
  Interventions: Other: Saline Solution (Control)

INTERVENTIONS:
Drug: 1: Vitamin C Supplementation — • Vitamin C (Ascorbic Acid): This intervention involves the administration of vitamin C, which is known for its antioxidant properties. The concentration will be 120 mg in 1.2 ml, and the produced volume will be divided by six lower anterior teeth; each tooth will receive 0.2 ml (20 mg) of the vitamin C. It is hypothesized to accelerate orthodontic tooth movement by reducing oxidative stress and promoting collagen synthesis.
  Arms: Arm 1: Vitamin C Treatment
Drug: Vitamin E Supplementation — • Vitamin E (Tocopherol Acetate): This intervention uses vitamin E, another antioxidant, thought to reduce inflammation and support tissue repair, potentially improving the effectiveness of orthodontic treatment by enhancing tissue recovery and reducing side effects. The concentration will be 60 mg in 0.4 ml, and the produced volume will be divided by six lower anterior teeth; each tooth will receive 0.07 ml (10 mg) of the vitamin E.
  Arms: Vitamin E Treatment
Other: Saline Solution (Control) — Saline Solution (Control): The control group will receive a saline solution, which is a placebo, allowing for the comparison of the effects of vitamin C and vitamin E on orthodontic tooth movement without the influence of additional nutrients.
  Arms: Arm 3: Saline Control

SUMMARY:
Brief Summary of the Study

This study investigates the effects of locally administered vitamins C and E on orthodontic tooth movement during the initial stage of treatment. Orthodontic tooth movement relies on bone remodeling, which can be influenced by antioxidants like vitamins C and E. Vitamin C promotes collagen formation and osteoblast activity, while vitamin E has anti-inflammatory and antioxidant properties that may impact bone metabolism.

The study is a randomized clinical trial conducted in multiple clinics, where patients will be divided into three groups:

1. Control group - receives a saline injection.
2. Vitamin C group - receives a local injection of vitamin C.
3. Vitamin E group - receives a local injection of vitamin E.

Injections will be administered every two weeks for six months, while patients undergo orthodontic treatment with fixed appliances. Researchers will evaluate the rate of tooth movement, root resorption, pain perception, and patient experience. Additionally, biomarkers related to bone remodeling will be measured in gingival crevicular fluid at different time points.

The study aims to determine whether local administration of vitamins C or E enhances orthodontic tooth movement and elevate their effects on the orthodontic potential side effects like root resorption and pain. The findings may provide valuable insights into optimizing orthodontic treatment with the help of antioxidants.

DETAILED DESCRIPTION:
This randomized clinical trial aims to investigate the effects of locally administered vitamins C and E on mandibular incisor crowding relief during the initial stage of orthodontic treatment. The study follows a multicenter, prospective, single-blinded, parallel-group design with equal randomization (1:1) and is conducted in private clinics and hospitals.

Study Rationale

Orthodontic tooth movement involves a complex biological process mediated by bone remodeling, which is regulated by mechanical forces and biochemical mediators. Oxidative stress and inflammatory responses play a significant role in the remodeling process. Vitamin C (ascorbic acid) and vitamin E (tocopherol) are known for their antioxidant properties and potential effects on bone metabolism, tissue healing, and inflammation modulation. This study aims to determine whether locally administered vitamins C and E can enhance orthodontic tooth movement, reduce adverse effects such as root resorption, and improve patient experience during treatment.

Study Objectives

The primary objective is to compare the effectiveness of vitamin C and vitamin E injections versus a saline control in mandibular incisor crowding relief over 24 weeks.

The secondary objectives include:

* Assessing the extent of apical root resorption using periapical radiographs.
* Evaluating pain perception using a Visual Analog Scale (VAS) during the first week after each archwire change.
* Measuring patient perception of treatment experience through a structured questionnaire.
* Analyzing levels of biomarkers associated with bone remodeling (RANKL, OPG, RUNX2) in gingival crevicular fluid (GCF) to determine the biological effects of the interventions.

Participant Selection

Eligible participants are patients aged 12 years and older with moderate to severe mandibular anterior crowding (Little's Irregularity Index [LII] of 4-9 mm). Exclusion criteria include systemic diseases, prior orthodontic treatment, or the use of medications that could influence bone metabolism or inflammatory responses.

Intervention Groups

Participants will be randomly assigned to one of three groups:

1. Control Group: Receives saline injection.
2. Vitamin C Group: Receives intraepidermal injection of vitamin C (120 mg in 1.2 ml, divided among six mandibular anterior teeth).
3. Vitamin E Group: Receives intraepidermal injection of vitamin E (60 mg in 0.4 ml, divided among six mandibular anterior teeth).

Injections are repeated biweekly for a total of six months (24 weeks).

Orthodontic Treatment Protocol

All participants undergo standardized orthodontic treatment using MBT brackets (0.022-inch slot). The leveling and alignment phase follows a sequential archwire progression with heat-activated nickel-titanium (HANT) archwires in the following sequence:

* 0.014-inch HANT (initial 4 weeks)
* 0.016-inch HANT (weeks 4-8)
* 0.018-inch HANT (weeks 8-24)

No additional orthodontic interventions, such as interproximal reduction or extractions, will be performed during the study period.

Data Collection and Outcome Assessments

Data will be collected at multiple time points throughout the study:

1. Mandibular Incisor Crowding Relief

   * 3D-scanned digital models will be used to measure Little's Irregularity Index (LII) at baseline and every 4 weeks until week 24.
2. Root Resorption

   * Standardized periapical radiographs of mandibular anterior teeth will be taken at baseline, 8 weeks, and 24 weeks to evaluate root resorption.
3. Pain Perception

   * Participants will record pain intensity on a VAS scale (0-10) during the first week after each wire change (every 4 weeks).
4. Patient Perception

   * A structured questionnaire assessing comfort, esthetics, and perceived treatment progress will be administered at 8 weeks.
5. Biomarker Analysis

   * Gingival crevicular fluid (GCF) samples will be collected at baseline, 1 week, and 4 weeks. Levels of RANKL, OPG, and RUNX2 will be analyzed to assess changes in bone remodeling activity.

Statistical Analysis

Data will be analyzed using SPSS v26.Statistical methods include:

* Descriptive statistics (mean, standard deviation, frequency).
* Reliability analysis for measurement consistency.
* Inferential statistics, including paired and independent t-tests, analysis of variance (ANOVA), and regression models, to compare treatment effects.

A significance level of 0.05 will be used for hypothesis testing.

Study Oversight and Ethical Considerations

The study is self-funded and complies with ethical guidelines for human research. Ethical approval is pending from the appropriate review board. All participants (or their legal guardians) will provide informed consent before enrollment.

Potential Impact

This trial may provide valuable insights into the role of antioxidant therapy in orthodontic treatment. If vitamins C and E positively influence tooth movement and root integrity, their use could enhance treatment efficiency while minimizing complications. Findings may also contribute to a better understanding of bone remodeling mechanisms in response to mechanical forces.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 12 years and above, who are indicated for fixed appliance orthodontic treatment.
2. Patients with moderate to severe crowding (4-9 mm) of the mandibular anterior teeth as per the Little's Irregularity Index (LII).
3. 4. Treatment with or without two mandibular first premolars extraction. Presence of all the mandibular permanent teeth, except the third molars.

5. The overbite and overjet should not impede bracket placement on the mandibular anterior teeth.

Exclusion Criteria:

1. History of previous orthodontic intervention.
2. History of trauma or root resorption in the mandibular anterior teeth.
3. Presence of mandibular anterior teeth crowding of less than 4 mm or greater than 9 mm (LII).
4. Existence of blocked-out teeth precluding engagement with the aligning archwire.
5. History of systemic diseases, especially diabetes and bone diseases.
6. Patients with periodontitis and obvious loss of tooth attachment according to Plaque and Bleeding on Probing indices.
7. Pregnant and lactating mothers.
8. Mouth breathing patients and smokers.
9. Healthy patients who have not used any medications (such as anti-inflammatory or antimicrobial drugs) or supplements (such as vitamins)

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-02-23 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Difference in the amount of crowding relief of the mandibular incisors before treatment and at 4, 8, 12, 16, 20, and 24 weeks after the start of treatment among the two vitamins and control groups | The amount of crowding relief will be measured using Little's Irregularity Index (LII) on 3D digital models of the mandibular anterior teeth. Measurements will be taken at baseline (T0) and at 4, 8, 12, 16, 20, and 24 weeks to assess changes over time.
  The amount of crowding relief will be measured using Little's Irregularity Index (LII) on 3D digital models of the mandibular anterior teeth. Pre-treatment (T0) and post-treatment models at 4, 8, 12, 16, 20, and 24 weeks will be compared.
  * Measurement method: Alginate impressions will be taken at each time point and converted into 3D digital models using a high-precision scanner.
  * Definition: LII quantifies anterior misalignment by summing the displacement between mesial and distal contact points of six mandibular incisors.
  * Units: Millimeters (mm), rounded to 0.01 mm.
  * Expected outcome: Greater LII reduction indicates a higher rate of tooth movement.
  * Comparison: The control (saline) group will be compared with the vitamin C and vitamin E groups to assess their effects on tooth movement.

SECONDARY OUTCOMES:
Pain Perception After Archwire Placement: A Visual Analog Scale Assessment | From the placement of each archwire to 7 days post-placement.
  Pain perception will be measured using a Visual Analog Scale (VAS), a commonly used tool in clinical settings to quantify subjective pain experiences. The VAS consists of a 10 cm line where participants mark their pain level. One end of the line represents "no pain" (score of 0), and the other end represents "worst pain imaginable" (score of 10). Participants will be asked to record their pain levels twice daily for the first 7 days following each archwire placement during the treatment phase.
Amount of orthodontically-induced inflammatory root resorption (OIIRR) in the apical region of mandibular anterior teeth | Pre-treatment (T0), 8 weeks (T1), and 24 weeks (T2) after the start of treatment.
  Measurement of the root resorption in the apical region of the mandibular anterior teeth, assessed through radiographs and calculated by comparing the root length and crown length.
Patient perception using a newly developed questionnaire for adjunctive orthodontic therapy | 8 weeks after the start of treatment.
  Patients will complete a questionnaire to assess their perception of the treatment's comfort, side effects, and any additional effects due to vitamin administration during orthodontic therapy.
Levels of biomarkers (RANKL, OPG, and RUNX2) in gingival crevicular fluid (GCF): | Pre-treatment (T0), 1 week (T1), and 4 weeks (T2) after the start of treatment.
  Measurement of the biomarkers in the GCF, which are involved in bone turnover and remodeling. These markers will help assess the biological effects of the vitamins on periodontal tissues during the initial stage of orthodontic treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Dr. Yassir Abdulkadhim Yassir, Ph.D. (Orthodontics) (UK), Study Director — University of Baghdad
Locations (3):
- Iraq (3):
  - Baghdad Al-Karkh Health Directorate, Baghdad, Iraq, Baghdad, Baghdad Governorate
  - Baghdad Al-Rusafa Health Directorate, Baghdad, Baghdad Governorate
  - College of Dentistry, University of Baghdad, Baghdad, Iraq, Baghdad, Baghdad Governorate

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bolat E, Esenlik E, Oncu M, Ozgocmen M, Avunduk MC, Yuksel O. Evaluation of the effects of vitamins C and E on experimental orthodontic tooth movement. J Dent Res Dent Clin Dent Prospects. 2020 Spring;14(2):131-137. doi: 10.34172/joddd.2020.0027. Epub 2020 Jun 17. PMID 32908655
- [Background] Yussif, N. (2019). Oral Mesotherapy: might be considered as an adjunctive technique for the different surgical procedures?. In Periodontal disease-diagnostic and adjunctive non-surgical considerations. IntechOpen.
- [Background] Yussif, N.M.A., Dehis, H.M., Rahman, A.R.A., Aziz, M.A.W.M.A. and Yassin, M.M. (2018). Efficacy and safety of locally injectable vitamin C on accelerating the orthodontic movement of maxillary canine impaction (oral mesotherapy technique): prospective study. Clinical Cases in Mineral & Bone Metabolism, 15(2).
- [Background] Mohsin MK, Qadir Omer Z. The effect of vitamin E incorporated into injectable platelet-rich fibrin on orthodontic tooth movement in rabbits. Cell Mol Biol (Noisy-le-grand). 2024 Jun 5;70(6):147-154. doi: 10.14715/cmb/2024.70.6.23. PMID 38836668
- [Background] Kappus H, Diplock AT. Tolerance and safety of vitamin E: a toxicological position report. Free Radic Biol Med. 1992;13(1):55-74. doi: 10.1016/0891-5849(92)90166-e. PMID 1628854
- [Background] Esenlik E, Naziroglu M, Acikalin C, Ovey IS. Vitamin E supplementation modulates gingival crevicular fluid lipid peroxidation and antioxidant levels in patients with orthodontic tooth movement. Cell Biochem Funct. 2012 Jul;30(5):376-81. doi: 10.1002/cbf.1833. Epub 2011 Nov 24. PMID 22113708
- [Background] Carr AC, Lykkesfeldt J. Discrepancies in global vitamin C recommendations: a review of RDA criteria and underlying health perspectives. Crit Rev Food Sci Nutr. 2021;61(5):742-755. doi: 10.1080/10408398.2020.1744513. Epub 2020 Mar 30. PMID 32223303
- [Background] Mucklow, J.C. (2000). Martindale: the complete drug reference. British journal of clinical pharmacology, 49(6), p.613.
- [Background] Hathcock JN, Azzi A, Blumberg J, Bray T, Dickinson A, Frei B, Jialal I, Johnston CS, Kelly FJ, Kraemer K, Packer L, Parthasarathy S, Sies H, Traber MG. Vitamins E and C are safe across a broad range of intakes. Am J Clin Nutr. 2005 Apr;81(4):736-45. doi: 10.1093/ajcn/81.4.736. PMID 15817846
- See also: Related Info — https://scholar.google.com/scholar?hl=en&as_sdt=0%2C5&q=Mucklow%2C+J.C.+%282000%29.+Martindale%3A+the+complete+drug+reference.+British+journal+of+clinical+pharmacology%2C+49%286%29%2C+p.613.+.+%3A+.+.&btnG=
- See also: Related Info — https://scholar.google.com/scholar?hl=en&as_sdt=0%2C5&q=Carr%2C+A.C.+and+Lykkesfeldt%2C+J.+%282021%29.+Discrepancies+in+global+vitamin+C+recommendations%3A+A+review+of+RDA+criteria+and+underlying+health+perspectives.+Critical+reviews+in+food+science+and+nutrition%2C+61%285%29%2C+pp.742-755.+&btnG=
- See also: Related Info — https://scholar.google.com/scholar?hl=en&as_sdt=0%2C5&q=Kappus%2C+H.+and+Diplock%2C+A.T.+%281992%29.+Tolerance+and+safety+of+vitamin+E%3A+a+toxicological+position+report.+Free+Radical+Biology+and+Medicine%2C+13%281%29%2C+pp.55-74.+.+%3A+.+.&btnG=
- See also: Related Info — https://scholar.google.com/scholar?hl=en&as_sdt=0%2C5&q=Esenlik%2C+E.%2C+Naz%C4%B1ro%C4%9Flu%2C+M.%2C+A%C3%A7%C4%B1kal%C4%B1n%2C+C.+and+%C3%96vey%2C+I.S.+%282012%29.+Vitamin+E+supplementation+modulates+gingival+crevicular+fluid+lipid+peroxidation+and+antioxidant+levels+in+patients+with+orthodontic+tooth+movement.+Cell+biochemistry+and+function%2C+30%285%29%2C+pp.376-381.+.+%3A+.+.&btnG=
- See also: Related Info — https://scholar.google.com/scholar?hl=en&as_sdt=0%2C5&q=Yussif%2C+N.M.A.%2C+Dehis%2C+H.M.%2C+Rahman%2C+A.R.A.%2C+Aziz%2C+M.A.W.M.A.+and+Yassin%2C+M.M.+%282018%29.+Efficacy+and+safety+of+locally+injectable+vitamin+C+on+accelerating+the+orthodontic+movement+of+maxillary+canine+impaction+%28oral+mesotherapy+technique%29%3A+prospective+study.+Clinical+Cases+in+Mineral+%26+Bone+Metabolism%2C+15%282%29.+.+%3A+.+.&btnG=
- See also: Related Info — https://scholar.google.com/scholar?hl=en&as_sdt=0%2C5&q=Yussif%2C+N.+%282019%29.+Oral+Mesotherapy%3A+might+be+considered+as+an+adjunctive+technique+for+the+different+surgical+procedures%3F.+In+Periodontal+disease-diagnostic+and+adjunctive+non-surgical+considerations.+IntechOpen.+.+%3A+.+.&btnG=
- See also: Related Info — https://scholar.google.com/scholar?hl=en&as_sdt=0%2C5&q=Mohsin%2C+M.K.+and+Omer%2C+Z.Q.+%282024%29.+The+effect+of+vitamin+E+incorporated+into+injectable+platelet-rich+fibrin+on+orthodontic+tooth+movement+in+rabbits.+Cellular+and+Molecular+Biology%2C+70%286%29%2C+pp.147-154.+.+%3A+.+.&btnG=
- See also: Related Info — https://scholar.google.com/scholar?hl=en&as_sdt=0%2C5&q=Bolat%2C+E.%2C+Esenlik%2C+E.%2C+%C3%96nc%C3%BC%2C+M.%2C+%C3%96zg%C3%B6%C3%A7men%2C+M.%2C+Avunduk%2C+M.C.+and+Y%C3%BCksel%2C+%C3%96.+%282020%29.+Evaluation+of+the+effects+of+vitamins+C+and+E+on+experimental+orthodontic+tooth+movement.+Journal+of+Dental+Research%2C+Dental+Clinics%2C+Dental+Prospects%2C+14%282%29%2C+p.131.+.+%3A+.+.&btnG=